CLINICAL TRIAL: NCT00981331
Title: Changes in the Ankle Range of Motion Following Subtalar Joint Manipulation in Patients With Sub-acute, Grade II, Ankle Inversion Sprains Quantified Using Quaternion Eigen Analysis.
Brief Title: Changes in the Ankle Range of Motion Following Subtalar Joint Manipulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators and resources are no longer available for completion of the study due to retirements, relocations and reassignments.
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Alex Lee, Clinician, Canadian Memorial Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 092025
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Ankle Inversion Sprain
Keywords: Subtalar joint; Musculoskeletal Manipulations; Manipulation, Chiropractic; Ankle sprain; Inversion sprain; Range of motion, Articular; Quaternion; Eigen analysis
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subtalar joint manipulation (Experimental): Each subject in this group will recieve a subtalar joint manipulation to their symptomatic ankle
  Interventions: Procedure: Subtalar joint manipulation
- Sham Manipulation (Sham Comparator): Each subject in this group will recieve a sham subtalar joint manipulation to their symptomatic ankle
  Interventions: Procedure: Sham subtalar joint manipulation

INTERVENTIONS:
Procedure: Subtalar joint manipulation — The intervention is defined as a toggle-recoil, high-velocity, low-amplitude subtalar joint manipulation.
  Other Names: Ankle manipulation
  Arms: Subtalar joint manipulation
Procedure: Sham subtalar joint manipulation — The sham manipulation is conducted by placing the ankle in a non-manipulative position, and the operator simply engages the toggle board to simulate the audible noise of the toggle board dropping. No force or thrust is applied to the ankle.
  Other Names: Sham manipulation
  Arms: Sham Manipulation

SUMMARY:
The purpose of the study is to determine whether manipulation of the subtalar joint (one of the two joints of the ankle) has an effect on ankle range of motion in a group of ankles that have sustained a subacute inversion ankle sprain.

The investigators expect subtalar joint manipulation will increase ankle range of motion about the subtalar joint, but not at the talocrural joint (the other joint of the ankle).

DETAILED DESCRIPTION:
Ankle inversion sprain is a common injury that can cause joint stiffness and range of motion deficits.(Holmer 1994, Beynnon 2001, Denegar 2002, Green 2001) Subtalar joint manipulation has been advocated as an intervention for inversion sprains to reduce pain, decrease joint stiffness, and improve range of motion.(Lopez-Rodriguez 2007)

The ankle is comprised of the talocrural and subtalar joints and their respective joint axes.(Hubbard 2006) Ankle rotation about these axes can be parameterized using quaternions, a four dimensional unit vector. Range of motion (ROM) about these axes can be determined by performing an eigen analysis of the quaternion matrices to determine the root mean squared values of the motion data about these axes.

The objective of the study is to investigate the immediate effects of subtalar joint manipulation on the ROM about the ankle's talocrural and subtalar joints on ankles that have sustained a subacute, grade II inversion sprain.

Forty patients with one sprained ankle and one asymptomatic ankle will be recruited. The subjects will be randomized into either a subtalar manipulation group or a sham manipulation group. The sprained ankle of each patient will receive either a standardized subtalar joint manipulation or a sham manipulation. The same patient's asymptomatic ankle will serve as the non-treatment control group. Range of motion pre- and post-manipulation will be quantified utilizing a quaternion eigen analysis. Kinematic and kinetic parameters will be collected during the manipulation to biomechanically characterize the manipulation. Pain pressure threshold and visual analog scale measurements for pain, stiffness, and quality of movement will be collected.

Our primary hypothesis is subtalar joint manipulation will increase subtalar ROM, but will have no effect on talocrural ROM. Our secondary hypothesis is subtalar joint manipulation will have positive effects on pain, stiffness, and quality of movement.

ELIGIBILITY:
Inclusion Criteria:

* Must have 1 ankle diagnosed with a subacute, grade II inversion ankle sprain and 1 asymptomatic ankle
* Pain on palpation of the medial subtalar joint line
* Manual restriction of subtalar eversion as assessed by a passive joint play test of subtalar joint mobility

Exclusion Criteria: (Pellow 2001, Fryer 2002, Lopez-Rodriguez 2007)

* Acute ankle or foot trauma occurring within 7 days of injury incident
* Acute or healing fracture
* Gross ligamentous mechanical instability (grade III ankle sprains)
* Syndesmosis injury
* Inflammatory arthritis
* History of previous medial ankle sprain
* Medial ankle instability
* Severely pronated feet determined by Foot Posture Index score > +9 (Redmond 2006)
* Connective tissue disorder (Grahame 2000)
* Benign joint hypermobility syndrome (Grahame 2000)

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Range of Motion determined by a biomechanical ankle model (quaternion eigen analysis) | Outcome measure will be collected immediately pre-manipulation and immediately post-manipulation on day of testing (ie. 1 day)

SECONDARY OUTCOMES:
Visual Analog Scales for self-reported pain, stiffness, and quality of movement | Outcome measure will be collected immediately pre-manipulation and immediately post-manipulation on the day of testing (ie. 1 day)
Pain pressure threshold | Outcome measure will be collected immediately pre-manipulation and immediately post-manipulation on the day of testing (ie. 1 day)
preload force | Outcome measure will be collected during the manipulation on the day of testing (ie. 1 day)
peak force | Outcome measure will be collected during the manipulation on the day of testing (ie. 1 day)
thrust duration | Outcome measure will be collected during the manipulation on the day of testing (ie. 1 day)
force - time slope | Outcome measure will be collected during the manipulation on the day of testing (ie. 1 day)
subtalar joint angle | Outcome measure will be collected during the manipulation on the day of testing (ie. 1 day)
talocrural joint angle | Outcome measure will be collected during the manipulation on the day of testing (ie. 1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander D Lee, BSc, DC, Principal Investigator — Canadian Memorial Chiropractic College; John J Triano, DC, PhD, Study Director — Canadian Memorial Chiropractic College
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Canadian Memorial Chiropractic College, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holmer P, Sondergaard L, Konradsen L, Nielsen PT, Jorgensen LN. Epidemiology of sprains in the lateral ankle and foot. Foot Ankle Int. 1994 Feb;15(2):72-4. doi: 10.1177/107110079401500204. PMID 7981804
- [Background] Beynnon BD, Renstrom PA, Alosa DM, Baumhauer JF, Vacek PM. Ankle ligament injury risk factors: a prospective study of college athletes. J Orthop Res. 2001 Mar;19(2):213-20. doi: 10.1016/S0736-0266(00)90004-4. PMID 11347693
- [Background] Denegar CR, Miller SJ 3rd. Can Chronic Ankle Instability Be Prevented? Rethinking Management of Lateral Ankle Sprains. J Athl Train. 2002 Dec;37(4):430-435. PMID 12937564
- [Background] Denegar CR, Hertel J, Fonseca J. The effect of lateral ankle sprain on dorsiflexion range of motion, posterior talar glide, and joint laxity. J Orthop Sports Phys Ther. 2002 Apr;32(4):166-73. doi: 10.2519/jospt.2002.32.4.166. PMID 11949665
- [Background] Green T, Refshauge K, Crosbie J, Adams R. A randomized controlled trial of a passive accessory joint mobilization on acute ankle inversion sprains. Phys Ther. 2001 Apr;81(4):984-94. PMID 11276181
- [Background] Lopez-Rodriguez S, Fernandez de-Las-Penas C, Alburquerque-Sendin F, Rodriguez-Blanco C, Palomeque-del-Cerro L. Immediate effects of manipulation of the talocrural joint on stabilometry and baropodometry in patients with ankle sprain. J Manipulative Physiol Ther. 2007 Mar-Apr;30(3):186-92. doi: 10.1016/j.jmpt.2007.01.011. PMID 17416272
- [Background] Hubbard TJ, Hertel J. Mechanical contributions to chronic lateral ankle instability. Sports Med. 2006;36(3):263-77. doi: 10.2165/00007256-200636030-00006. PMID 16526836
- [Background] Pellow JE, Brantingham JW. The efficacy of adjusting the ankle in the treatment of subacute and chronic grade I and grade II ankle inversion sprains. J Manipulative Physiol Ther. 2001 Jan;24(1):17-24. doi: 10.1067/mmt.2001.112015. PMID 11174691
- [Background] Fryer GA, Mudge JM, McLaughlin PA. The effect of talocrural joint manipulation on range of motion at the ankle. J Manipulative Physiol Ther. 2002 Jul-Aug;25(6):384-90. doi: 10.1067/mmt.2002.126129. PMID 12183696
- [Background] Grahame R, Bird HA, Child A. The revised (Brighton 1998) criteria for the diagnosis of benign joint hypermobility syndrome (BJHS). J Rheumatol. 2000 Jul;27(7):1777-9. No abstract available. PMID 10914867
- [Background] Redmond AC, Crosbie J, Ouvrier RA. Development and validation of a novel rating system for scoring standing foot posture: the Foot Posture Index. Clin Biomech (Bristol). 2006 Jan;21(1):89-98. doi: 10.1016/j.clinbiomech.2005.08.002. Epub 2005 Sep 21. PMID 16182419